CLINICAL TRIAL: NCT00621426
Title: T-Wave Alternans in Dialysis Patients
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: General Electric (Industry)
Responsible Party: Principal Investigator, Rod Passman, Principal Investigator, Northwestern University
Other Study IDs: 0388-010
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Sudden Cardiac Death; End Stage Renal Disease
Keywords: T wave alternans (TWA); dialysis; end stage renal disease; sudden cardiac death; T-wave alternans; Cardiac electrical instability; Sympathetic and electrolyte-induced alterations; Ventricular repolarization
MeSH Terms: conditions — Death, Sudden, Cardiac; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Patients with end-stage renal disease (ESRD) treated with hemodialysis three (3) times per week for at least 3 continuous months

SUMMARY:
Sudden cardiac death due to arrhythmia is the leading cause of death in end-stage renal disease (ESRD) patients treated with hemodialysis (HD). As it is anticipated that the number of individuals with ESRD will exceed 1.2 million in the next 20 years, sudden death in this population has enormous public health impact. Research has shown that arrhythmic events are temporally associated with longer periods between HD with a three-fold risk of events in the 12 hours preceding the longest inter-dialysis interval. The exact cause of these findings is unknown.

DETAILED DESCRIPTION:
The purpose of this study is to assess the degree of cardiac electrical instability at various times in the dialysis cycle. The hypothesis is that longer time intervals between hemodialysis results in sympathetic and electrolyte-induced alterations in ventricular repolarization that can be measured non-invasively using microvolt T-wave alternans (TWA). This increase in cardiac electrical instability may serve as a link between the clinically observed periods of increased risk and the occurrence of sudden cardiac death.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic ESRD who have been on HD for at least 3 months
* Subjects 18 to 90 years of age with one or more risk factors for coronary artery disease or sudden cardiac death, including diabetes, peripheral vascular disease, known coronary artery disease, or ejection fraction < 40% by any imaging modality.

Exclusion Criteria:

* Subjects unwilling or unable to give written informed consent.
* Patients unable to return for regularly scheduled dialysis treatments
* Atrial fibrillation or flutter at screening
* Major surgical procedure two months prior to enrollment
* High grade heart block or a permanent pacemaker in situ
* Patients with known allergies to adhesive tape

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end-stage renal disease (ESRD) treated with hemodialysis three (3) times per week for at least 3 continuous months will be enrolled. No limitations for gender, race, socioeconomic status or any other parameters will be applied.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Measure the degree of cardiac electrical instability at various times in the dialysis cycle. | Basline, during dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Rod Passman, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States